CLINICAL TRIAL: NCT07014605
Title: Implementing Sustainable Mobile Health Technology to Optimize Smoking Cessation Program for Lao People With HIV
Brief Title: Smoking Cessation Program for Lao People With HIV
Acronym: I-STOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Laboratory and Epidemiology, Lao PDR (Other); National Tobacco Control Committee, Lao PDR (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 17386; U01CA294811 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation; HIV
Keywords: smoking cessation; cancer control; implementation science; low- and middle-income countries; mobile health
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA-SH (Ask-Advise-Connect paired with self-help material) (Active Comparator): Participants will receive advice to quit smoking and be provided with a self-help guide to support smoking cessation.
  Interventions: Behavioral: Smoking Cessation Self Help Guide
- AA-MAP (Ask-Advise-Connect paired with mHealth-based automated treatment program) (Experimental): Participants will receive advice to quit smoking and be connected to the mHealth-based automated treatment program (MAP). MAP is a fully automated smartphone-based treatment program that involves interactive and personalized proactive messages, images, or videos.
  Interventions: Behavioral: Smartphone-delivered Automated Messaging

INTERVENTIONS:
Behavioral: Smoking Cessation Self Help Guide — Our team has translated and validated the World Health Organization's "A guide for tobacco users to quit" into Lao language for use as the self-help guide in this study. Attached to the guide is an information sheet regarding NRT (e.g., patches and lozenges), where to buy them, and how to use them.
  Arms: AA-SH (Ask-Advise-Connect paired with self-help material)
Behavioral: Smartphone-delivered Automated Messaging — The MAP includes text messages, images, and videos with content designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The MAP will begin immediately after enrollment and continue for a 26-week period. The MAP approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
  Arms: AA-MAP (Ask-Advise-Connect paired with mHealth-based automated treatment program)

SUMMARY:
Tobacco use remains the leading modifiable risk factor for preventing cancer globally, particularly among people with HIV (PWH). In Laos, 61-80% of male PWH and 3-10% of female PWH smoke cigarettes. PWH who smoke in Laos have no reliable smoking cessation support. Thus, implementing sustainable and evidence-based smoking cessation interventions for PWH in Laos is needed. The investigators developed a scalable and affordable mHealth-based automated treatment program (MAP) to support Lao and Cambodian smokers to quit smoking. MAP involves interactive, tailored, personalized content (text messages, photos, and videos) delivered via a smartphone app. Along with effective cessation treatments, it is imperative to implement procedures to identify patients who smoke and to connect them to treatment. Our team pioneered the Ask-Advise-Connect (AAC, asking patients about smoking at every visit, briefly advising those who smoke to quit, and connecting them to treatment) approach, which showed great impact in our previous US studies. The purpose of this study is to compare 2 smoking cessation implementation strategies in 8 antiretroviral therapy (ART) clinics in the 6 most populous regions in Laos, using a hybrid type-2 pragmatic effectiveness-implementation study and a parallel cluster randomized trial design. Specifically, the investigators will compare an AAC approach paired with our previously developed MAP (AA-MAP) to an AAC approach paired with less resource-intensive printed self-help material (AA-SH). The investigators will use the Practical, Robust Implementation and Sustainability Model (PRISM), which expands the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework to include more contextual factors relevant to program implementation. Aim 1 is to evaluate the reach and effectiveness of AA-MAP versus AA-SH. Reach is the proportion of PWH who smoke and are willing to make a quit attempt that enroll in treatment. Effectiveness is the proportion of enrolled participants who achieve biochemically confirmed point prevalence abstinence 6 months after enrollment. The investigators will also estimate the real-world impact (impact = reach × effectiveness) of each intervention. Aim 2 is to determine other implementation outcomes of AA-MAP and AA-SH. Aim 3 is to assess the resource use and costs of implementing AA-MAP and AA-SH. The project has the potential to transform HIV care and to reduce tobacco-related cancers and other morbidities.

DETAILED DESCRIPTION:
Experimental Design: The investigators chose cluster (vs. individual) randomized controlled trial (RCT) design as it is a robust, pragmatic design for service interventions (AA-SH/AA-MAP) at the cluster (ART clinics) level rather than the patient level. They considered a stepped-wedge design, which would have allowed all clinics to receive both interventions during the trial and within-cluster comparisons. However, that would have presented the risk of unequal chronological exposure to interventions, and the potential risk of internal contamination due to carry-over effects (i.e., during the 6-month treatment period, enrollees may be exposed to the other intervention if the clinic switched interventions). Thus, the investigators chose the parallel cluster RCT design but will allow all clinics the option to implement both AA-SH and AA-MAP after the trial period.

Study sites and participant recruitment: Participants will be recruited from 8 ART clinics in the 6 provinces/regions that are most populous or have an increasing HIV+ incidence. Besides currently registered patients, these clinics together gain approximately 1,500 new patients each year. These clinics provide comprehensive care for registered ART patients, including ART, ART adherence counseling, nutrition, risk-reduction counseling, and treatments for comorbidities other than tobacco use. Registered patients have periodic prescheduled appointments (about once per month for new patients and once per 4 months for patients with controlled viral load). To avoid potential skewness, the investigators will create 2 sets of 4 clinics with comparable patient populations and available resources and then randomly assign each set to an implementation strategy (AA-SH or AA-MAP).

Evaluation of reach and effectiveness of the AA-SH/AA-MAP approaches: In clinics assigned to AA-SH, staff will ask the patient if s/he smokes at every visit, advise smokers to quit, ask if they want to receive help with quitting, and provide them with a self-help guide. The AA-SH will be performed by counselors (counseling sessions occur at almost every visit and counselors have more time with patients) or nurses (when vital signs or blood samples are collected). It is optional for physicians to provide additional brief advice to quit (physicians have a more authoritative voice in Asian culture but less time with patients). The investigators will document which types of healthcare professionals provide advice to quit for additional analysis. The clinic staff will use a short form attached to patients' paper medical records to perform AA-SH, with a standardized question about smoking status (Did you [participant] smoke cigarettes in the past 7 days? [Yes/No]), a sample script to briefly advise smokers to quit, and 2 standardized questions about intent to quit (Are you [participant] willing to make a quit attempt in the next 2 weeks? [Yes/Remind me later], and if yes: Do you [participant] want to receive more information regarding how to quit? [Yes/No]). Those who answer yes to both questions will be provided with the self-help guide. The staff will also ask patients if they consent to be contacted at 6 months by research staff. The self-help guide is a 22-page booklet that the investigators developed in our R21/R33 study. Attached to the guide is an information sheet regarding NRT (e.g., patches and lozenges), where to buy them, and how to use them. On a weekly basis, clinic staff enter patients' new information collected via paper medical records into DHIS2 database. At this time, clinic staff will also enter the data collected for this study into DHIS2 database.

In the AA-MAP arm, clinic staff will do the ask-advise steps, and then will ask if smokers use a smartphone and proactively connect them to the MAP. Specifically, clinic staff will show a QR code (linked to a brief REDCap form) to smokers, and guide them through scanning the QR code, answering the few questions on the landing page (about their names and contact information), and submitting the form. Through our ongoing studies in Laos, NCLE/NTCC staff members have been proficient at managing the mHealth platform and app; these will serve in the MAP core team to provide technical assistance to all end users. Within 48 hours of receiving the REDCap form, MAP core staff will communicate with the enrollees to instruct them to download, sign up, and use the smoking cessation app. An instructional video of these steps will also be sent to the enrollees. For smokers who do not have a smartphone, the clinic staff will explain that the smoking cessation intervention will be available to them in the future. Our smoking cessation app is fully automated and interactive. Its content is adapted from the team's previous efforts and from the WHO/US NCI-suggested message banks. MAP is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills and social support, and to reduce nicotine withdrawal symptoms and stress. The mHealth treatment will begin immediately after enrollment and will continue for 26 weeks. MAP allows for several levels of personalization and tailoring for each participant. First, at Day 1, participants will be asked some questions about their biological sex, past quit attempts, and the presence or fear of specific comorbidities. Messages tailored to these responses will be delivered automatically throughout the treatment period. Second, there will be different bins of messages for different cessation phases to ensure that the intervention content targets critical mechanisms of each phase. Phase identification follows the PBM's suggestion: preparation (enrollment to quit date), cessation (quit date to 4 weeks post-quit date), and maintenance (4-26 weeks post-quit date). Finally, the app will prompt participants to complete a brief (4-6 items) assessment every week (e.g., stress or self-efficacy levels); answers to these questions will drive the delivery of appropriate content to each participant.

Training ART clinic staff: All potential AAC implementers at each ART clinic will receive an initial 2-hour in-person group training on implementing AAC and documenting data in the DHIS2 system. The training also includes information on why PWH should quit smoking, the effectiveness of the AAC approach in high-income countries, healthcare provider roles, available NRTs in Laos, and time for questions and answers. The initial training will be held immediately prior to the launch of the AA-SH/AA-MAP implementation at the ART clinics and will emphasize the importance of fidelity to AA-SH/AA-MAP. The initial training will be video recorded for future review and for training of newly hired clinic staff. There will be 4 "booster" training sessions at months 1, 6, 12, and 18 to reinforce the information in the initial training, address emerging issues, and answer clinic staff's questions. These 30-minute booster sessions will coincide with required clinic-wide staff meetings. Both the initial and booster training sessions will involve didactic lectures and role-playing exercises.

Other strategies to ensure treatment and implementation fidelity: The investigators will also use other strategies as recommended by the NIH Behavior Change Consortium and Carroll's conceptual framework for implementation fidelity to maximize fidelity across multiple clinics. These include all clinics following a standardized protocol, building the standardized AAC component into the medical questionnaire and DIHS2 platform, and monitoring AA-SH/AA-MAP enrollment in the DIHS2 database.

Assessment of reach and effectiveness. PWH who smoke and are willing to make a quit attempt within the next 2 weeks will be offered treatment (self-help guide or MAP). Reach is the proportion who enroll in treatment. The pool of participants for the assessment of effectiveness is AA-SH/AA-MAP enrollees. At 6 months post-enrollment, the research team will assess the smoking status of enrollees through a survey. Participants who self-report quitting will be seen in person at the clinic within 30 days post-survey for biochemical verification. The investigators will try to arrange this visit to coincide with participants' regular/prescheduled clinic visit for ART or other services. A local research staff member (not associated with ART clinics) will collect the data using the REDCap mobile app on a tablet. The research staff will assess up to 1,200 treatment enrollees at 6 months.

Other outcomes: The investigators will also estimate the impact of AA-SH and AA-MAP. Impact, the multiplicative effect of reach and effectiveness, is crucial in evaluating health intervention implementation. An intervention may have a broad reach but limited effectiveness, or have strong effectiveness but limited reach, and hence ultimately may have limited public health impact.

Evaluation of other multi-level implementation outcomes of AA-SH/AA-MAP: The investigators will use a mixed methods approach to assess other PRISM-based implementation outcomes (e.g., adoption, implementation fidelity, and sustainability) and to identify key determinants associated with these outcomes (e.g., intervention characteristics, patient characteristics, organization characteristics, or external factors). The investigators will use the convergent mixed methods design, in which quantitative and qualitative data are collected separately and then merged in analysis for interpretation.

Evaluation of the resource/cost associated with AA-SH/AA-MAP: To inform the decision-making of public sector stakeholders, the investigators will conduct an assessment of the resources needed to widely implement the interventions, and the potential gain from investing those resources from the perspective of the governmental service-providers.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years
2. reachable within 30 days of the target assessment date by different methods (up to 4 phone calls at different days and time, 3 text messages for each platform [e.g., SMS, Telegram, or Whatsapp], 3 emails if applicable, and via direct contact at a prescheduled clinic appointment if applicable)
3. consenting to be contacted after 6 months at the enrollment and able to provide recorded verbal informed consent when contacted by the research staff to participate.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Reach | At the end of the AA-SH/AA-MAP implementation at each ART clinic (up to 30 months)
  Reach is the proportion of PWH who smoke and are willing to make a quit attempt that enroll in treatment.
Effectiveness | 6 months post enrollment
  Effectiveness is the proportion of enrolled participants who achieve biochemically confirmed point prevalence abstinence 6 months after enrollment. Abstinence will be defined as biochemically confirmed self-reported 7-day point prevalence abstinence with expired CO <6 ppm.

SECONDARY OUTCOMES:
Impact | At the end of the individual and clinic data collection (up to 36 months after the start of the AA-SH/AA-MAP implementation)
  Impact = reach × effectiveness of each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Phonepadith Xangsayarath, MD, PhD, Study Director — Ministry of Health of Lao PDR, National Center for Laboratory and Epidemiology; Cate Moriasi, PhD, Study Director — The University of Oklahoma Health Sciences Center (OUHSC)
Locations (1):
- Setthathirath Hospital, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared upon request, with an established data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After data collection is complete.
Access Criteria: After an institutionally approved data sharing agreement is established, deidentified IPD will be shared via a secure data transfer mechanism approved by OUHSC. Data sharing requests will be reviewed and approved by the PI and OUHSC.